CLINICAL TRIAL: NCT06388174
Title: Idiopathic Generalized Epilepsy Syndromes: Clinical Features and Long-term Outcomes
Brief Title: Idiopathic Generalized Epilepsy Syndromes
Status: Recruiting | Type: Observational
Sponsor: Shen Chun-Hong (Other)
Responsible Party: Sponsor-Investigator, Shen Chun-Hong, Associate Senior Doctor, Second Affiliated Hospital, School of Medicine, Zhejiang University
Organization: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Other Study IDs: S2022-0336
Record Dates: First submitted 2024-04-16; First posted 2024-04-29 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy; Epilepsy, Idiopathic Generalized
MeSH Terms: conditions — Epilepsy; Epilepsy, Idiopathic Generalized

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
The idiopathic generalized epilepsies (IGEs) have historically included the syndromes childhood absence epilepsy (CAE), juvenile absence epilepsy (JAE), juvenile myoclonic epilepsy (JME), and epilepsy with generalized tonic-clonic seizures alone (GTCA). Recognition of the IGEs is important for clinical care, as it informs diagnosis, prevents unnecessary investigation, allows optimal selection of anti-seizure medications (ASMs), and provides prognostic guidance.

According to the new ILAE definition in 2022, the study aims to describe the clinical features, electroencephalographic, imaging findings and long-term prognosis.

DETAILED DESCRIPTION:
the Long-term prognosis include the rate of drug-resistent epilepsy, relapse after drug withdrawn, common comorbidities such as mood disorders, attention deficit hyperactivity disorder (ADHD) and learning disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Patients are consecutively and prospectively enrolled from epilepsy center, with newly diagnosed epilepsy or established epilepsy.
* Patients have a diagnosis of idiopathic generalized epilepsy (IGE), according to the 2022 diagnostic criteria.
* Comprehensive clinical information is collected, and 24 hour video-electroencephalography is performed.
* Sign the informed consent forms.

Exclusion Criteria:

* Other epilepsy syndromes are considered during follow-up, such as genetic generalized epilepsy.
* Lost to follow-up

Ages: 4 Years to 40 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients are consecutively and prospectively recruited from epilepsy center and clinics
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of drug-resistent epilepsy | through study completion, an average of 1 year
  We defined drug-resistant cases as those patients who have failed two or more trials of broad-spectrum ASMs or those otherwise indicated in IGE syndromes
The proportion of seizure freedom | through study completion, an average of 1 year
  We defined seizure freedom according to the International League Against Epilepsy (ILAE) definition

SECONDARY OUTCOMES:
The proportion of psychiatric comorbidity | through study completion, an average of 1 year
  The psychiatric comorbidities mainly include anxiety and depression, which are evaluated by Hamilton anxiety scale and Hamilton depression scale, respectively.
The proportion of psychosocial outcome | through study completion, an average of 1 year
  such as university entrance, marry
The proportion of seizure relapse after antiseizure medication withdrawn | through study completion, an average of 1 year
  Antiseizure medication withdrawn should be recommended by epilepsy experts

CONTACTS AND LOCATIONS:
Overall Officials: Chunhong Shen, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No